CLINICAL TRIAL: NCT02671656
Title: Reliability Assessment of the HumaSens Plus Measurement of Uricemia in Capillary Blood
Brief Title: Study of the Reliability of a Device (HumanSens Plus) Allowing Immediate Measurement Uric Acid in the Blood Obtained by Finger Tip Puncture.
Acronym: URICA
Status: Withdrawn | Type: Observational
Why Stopped: faisability
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ART-Viggo, Rheumatology department, Lariboisière Hospital, Paris, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: UC1501
Record Dates: First submitted 2016-01-29; First posted 2016-02-02 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Diabetes
Keywords: Uricemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperuricemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Uricemia — serum uric acid levels is measured once from venous blood samples in the biochemistry laboratory using standard automated colorimetric methods

SUMMARY:
Lowering the level of uric acid in the serum under 6mg/dL on the long term is a key factor of gout management success. Monitoring of uricemia in gout patients is therefore important and is presently done in the laboratory on serum samples obtained after venous puncture. This study aims at assessing the reliability of immediate uricemia measurement in a blood sample obtained by a mere fingertip puncture, by the HumaSensplus system, which is commercially available in the EU. Results obtained by the Humasens device will be compared to those of the standard measurement technique in serum and with a reference technique (liquid chromatography and mass spectroscopy). If the device appears reliable, it will allow self-measurement of uric acid by the gouty patient, in a similar way as diabetic patients measure their glycaemia following a fingertip puncture. This should improve patient monitoring and management effects.

DETAILED DESCRIPTION:
The aim of this study is

* to assess the validity of the capillary measure of uric acid level by the HumaSens plus system by comparing the measurement of total blood uric acid level by the HumaSens plus system with the routine measurement of serum uric acid by a standard and validated automated colorimetric method (primary objective).
* to look for a systematic bias and confounding factors (secondary objectives)

Methods

Design : This is a mono-centric prospective study. Patients will be recruited from the diabetology day hospital of hospital Lariboisière, Paris

Data collection : For each patient included at the Lariboisière Diabetology day hospital and included in this study, serum uric acid levels will be measured once from venous blood samples in the biochemistry laboratory using standard automated colorimetric methods, as presently routinely done and by liquid chromatography coupled with mass spectroscopy. In, addition, uric acid levels will also be simultaneously measured from capillary blood with the HumaSensplus system.

Hematocrit, glucose, cholesterol and triglycerides will be measured as well from venous blood samples and taken medications will be listed.

Planned analysis :

Planned sample size:

To obtain an estimated intraclass correlation of 0,800, with a two-sided 95% confidence interval with a width of 0,100, if the uric acid level is measured twice for each subject, we calculated that we needed a random sample of 204 subjects.

Statistical analyses:

Primary aim This study aims at studying the reliability of measurements of acid uric level by HumanSensplus against laboratory and measurements by liquid chromatography coupled with mass spectroscopy on serum from venous blood. There is no structure to the replicate measurements in the sense that nothing ties the first or second measurement on one patient to the first or second on another. The study thus conforms to a one-way random effect model. The data will be analyzed using a one-way random-effects ANOVA model.

The estimator of the intraclass correlation coefficient will be

With BMS=between-subject mean square, WMS=within-subject mean square and k0 = number of replicates. In this study k0=2.

The intraclass correlation coefficient will be calculated and the two-sided 95%CI will be provided for each comparison.

In addition differences between measurements will be plotted against mean of measurements in accordance with Bland and Altman.

Secondary aims The search for systematic bias and effect of confounding factors (hematocrit, glycemia, lipid concentrations and concomitant medications) will use different models of multiple regression

Logistic aspects

Ethical aspects:

Agreement will be sought from the local Ethics committee. All patients will be fully informed and will be provided with an information form. The data will be entered into an excel database and will be analysed anonymously. Fingertip glycaemia is presently systematically obtained in all these day hospital patients, and the addition of fingertip uricaemia in view of substituting this measurement to the systematic serum uric acid measurement presently done from a venous system in the biochemistry laboratory can be considered as a mere attempt to improve routine patient care.

Inclusion procedure:

The study will target 200 patients seen in diabetology day hospitalisation and fulfilling the inclusion criteria. As 15 patients are seen in the diabetology day hospitalisation ward every day, we estimate that the necessary patients sample size could be obtained within 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in the diabetology day hospital
* Patients aged at least 18 years-old
* French-speaking patients
* Patients able to understand the study and the information form

Exclusion Criteria:

* Patients unable to understand the aim of study aind the information sheet
* Patients not affiliated to a social security scheme (beneficiary or assignee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Uricemia | Day0
  Comparison the measurement of uric acid level by the HumaSensplus system with the routine measurement of uric acid by the automated colorimetric uricase method (Abbot), and with a reference method: liquid chromatography coupled with mass spectroscopy.
  This will be done once for every patient.

SECONDARY OUTCOMES:
Uricemia on capillary blood vs on serum | Day0
  Search for a systematic bias (the HumaSens measurement is on capillary blood whereas the other techniques are done on serum)
Haematocrit, glucose and lipid levels, medications | Day0
  Search for confounding factors (haematocrit, glucose and lipid levels, medications) which may affect the results of the HumaSens measurement

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BARDIN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Rhumatologie, Hôpital Lariboisière, Paris, France

IPD SHARING:
Plan to Share IPD: No